CLINICAL TRIAL: NCT00229216
Title: A Phase III Randomized, Multi-center, Double-blind, Double-dummy, Placebo-controlled Treatment Trial of Bacterial Vaginosis With Tinidazole Oral Tablets.
Brief Title: Treatment of Bacterial Vaginosis With Oral Tinidazole
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mission Pharmacal (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: T-500
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Bacterial Vaginosis
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — Tinidazole

INTERVENTIONS:
Drug: Tinidazole

SUMMARY:
The purpose of this study is to confirm the safety and efficacy of oral tinidazole for the treatment of bacterial vaginosis.

DETAILED DESCRIPTION:
Tinidazole is a second-generation nitroimidazole i.e. an updated form of the standard drug used to treat bacterial vaginosis (metronidazole). Two dosing regimens are being compared to placebo to treat bacterial vaginosis, one of the most common vaginal infections.

ELIGIBILITY:
Inclusion Criteria:

Clinical and microbiological diagnosis of bacterial vaginosis -

Exclusion Criteria:

Other sexually transmitted disease

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2005-01; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Therapeutic efficacy
Safety

SECONDARY OUTCOMES:
Clinical efficacy
Microbiological efficacy

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University School of Medicine, Durham, North Carolina, United States

REFERENCES:
- [Derived] Livengood CH 3rd, Ferris DG, Wiesenfeld HC, Hillier SL, Soper DE, Nyirjesy P, Marrazzo J, Chatwani A, Fine P, Sobel J, Taylor SN, Wood L, Kanalas JJ. Effectiveness of two tinidazole regimens in treatment of bacterial vaginosis: a randomized controlled trial. Obstet Gynecol. 2007 Aug;110(2 Pt 1):302-9. doi: 10.1097/01.AOG.0000275282.60506.3d. PMID 17666604